CLINICAL TRIAL: NCT05229796
Title: Pharmacokinetics and Bioequivalence of Two Empagliflozin, With Evaluation in Healthy Jordanian Subjects Under Fasting and Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mutah University (Other)
Responsible Party: Principal Investigator, Wael Abu Dayyih, Professor, Mutah University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 17-2021-SRES-4
Record Dates: First submitted 2022-01-18; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-01

CONDITIONS: Pharmacokinetic Parameters
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting state (Active Comparator)
  Interventions: Drug: Empagliflozin 10 mg Tab
- Fed state (Active Comparator)
  Interventions: Drug: Empagliflozin 10 mg Tab

INTERVENTIONS:
Drug: Empagliflozin 10 mg Tab — The Empagliflozin 10 mg Tab were administered orally. The plasma concentrations of empagliflozin were determined using an HPLC-MS/MS method. Tolerability and safety were assessed throughout the study. This study included 26 subjects, 26 in each fasting and fed group.

SUMMARY:
Background: The current study is a randomized, open-label, two-period, two-sequence, two-way crossover pharmacokinetic study in healthy Jordanian subjects to evaluate the pharmacokinetics and bioequivalence profile of two formulations of empagliflozin 10-mg under fasting and fed conditions administered orally.; (2) Methods: The plasma concentrations of empagliflozin were determined using High-performance liquid chromatography- Mass Spectrometry/ Mass Spectrometry (HPLC-MS/MS) method. This study included 26 subjects, 26 in each fasting and fed group.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

* healthy
* Jordanian volunteers
* some private hospitals (Amman, Jordan) Phase I Clinical Unit

Exclusion Criteria:

* Smokers
* heavy drinkers
* those who used CYP enzyme inhibitors within the previous 60 days
* those who had taken any medicine within the previous four weeks
* those who had a history of medication allergies
* those who had participated in previous clinical studies within the previous six months
* those with any significant clinical abnormality

Ages: 25 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2021-05-17 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
The plasma concentrations of empagliflozin were determined using an HPLC-MS/MS method. | 5 months
  The plasma concentration of empagliflozin under fasting and fed conditions states were measured using HPLC-MS/MS method and recorded in nmol\L.

CONTACTS AND LOCATIONS:
Locations (1):
- Wael Abu Dayyih, Amman, None Selected, Jordan

IPD SHARING:
Plan to Share IPD: Undecided